CLINICAL TRIAL: NCT07107256
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Phase III Clinical Trial to Evaluate the Efficacy and Safety of TQC2731 Injection in Patients With Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)
Brief Title: Clinical Trial of TQC2731 Injection in Patients With Chronic Sinusitis and Nasal Polyps
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Chia Tai Tianqing Pharmaceutical Technology Development Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQC2731-III-02
Record Dates: First submitted 2025-07-23; First posted 2025-08-06 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-04

CONDITIONS: Chronic Rhinosinusitis With Nasal Polyps (CRSwNP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQC2731 injection (Active Comparator): TQC2731 injection/placebo，4 weeks as a treatment cycle.
  Interventions: Drug: TQC2731 injection
- Placebo of TQC2731 (Placebo Comparator): TQC2731 injection/placebo，4 weeks as a treatment cycle.
  Interventions: Drug: Placebo of TQC2731

INTERVENTIONS:
Drug: TQC2731 injection — TQC2731 injection is a humanized monoclonal antibody that targets TSLP, blocks the TSLP signaling pathway, inhibits the production of downstream cytokines, and exerts anti-inflammatory effects.
  Arms: TQC2731 injection
Drug: Placebo of TQC2731 — TQC2731 injection is a humanized monoclonal antibody that targets TSLP, blocks the TSLP signaling pathway, inhibits the production of downstream cytokines, and exerts anti-inflammatory effects.
  Arms: Placebo of TQC2731

SUMMARY:
TQC2731 injection is a humanized monoclonal antibody that targets Thymic Stromal Lymphopoietin (TSLP), blocks the TSLP pathway, and inhibits the production of downstream cytokines, thereby exerting anti-inflammatory effects. The purpose of this study is to evaluate the efficacy and safety of TQC2731 injection in patients with chronic rhinosinusitis with nasal polyps (CRSwNP).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form prior to trial participation, demonstrating full understanding of trial objectives, procedures, and potential adverse reactions.
* Age between 18 and 75 years (inclusive) at the time of informed consent signing, regardless of gender.
* Diagnosis of bilateral chronic rhinosinusitis with nasal polyps (CRSwNP) meeting the diagnostic criteria of the "Chinese Guidelines for the Diagnosis and Treatment of Chronic Rhinosinusitis (2018)"
* At least one prior course of systemic corticosteroids (prednisone 0.5-1 mg/kg/day or 15-30 mg/day or equivalent for minimum 5 days) within 2 years before screening, with persistent bilateral CRSwNP; AND/OR contraindication/intolerance to systemic corticosteroids; AND/OR prior nasal polyp surgery performed more than 6 months before screening.
* Bilateral Nasal Polyp Score (NPS) ≥5 (maximum score 8) with ≥2 points per nostril, as assessed by nasal endoscopy during screening and randomization.
* Nasal Congestion Score (NCS) ≥2 at screening (daily average) and randomization (weekly average).
* Persistent symptoms of rhinorrhea and/or hyposmia/anosmia for over 8 weeks prior to screening.
* 22-item Sino-Nasal Outcome Test (SNOT-22) score ≥30 at screening and randomization.
* Stable dose of intranasal corticosteroids (INCS) for >4 weeks prior to screening (subjects using non-mometasone furoate nasal spray [MFNS] products must agree to switch to Mometasone Furoate Nasal Spray (MFNS) during the study).
* Subjects with comorbid asthma must have had stable asthma symptoms for ≥4 weeks prior to screening (if using medications, such as inhaled corticosteroids, the same dose must have been stably maintained for ≥4 weeks before screening, and the dose is assessed to remain stable during the first phase).
* The evaluation during the lead-in period showed that the medication adherence to intranasal mometasone furoate nasal spray (MFNS) was greater than 70%, and the adherence to daily symptom assessment records in the subjects' electronic logs was also greater than 70%. Note: Days with missing electronic log data were considered non-adherent to this criterion.
* Agreement to practice effective non-pharmacologic contraception from informed consent until 6 months post-final dose, for subjects/partners of childbearing potential.

Exclusion Criteria:

* Conditions/Diseases Affecting Efficacy Evaluation

  * Nasal septum deviation causing ≥1 nostril obstruction；
  * Perforation of the nasal septum
  * Acute sinusitis, nasal infection, or upper respiratory infection within 2 weeks pre-screening or during screening/run-in periods；
  * Rhinitis medicamentosa；
  * Eosinophilic granulomatosis with polyangiitis (EGPA), granulomatosis with polyangiitis (GPA), Young's syndrome, Kartagener's syndrome, other ciliary dyskinesia syndromes, or cystic fibrosis；
  * Suspected or confirmed fungal sinusitis by imaging；
  * Prior nasal surgery altering lateral wall structure precluding NPS assessment；
  * Nasal malignancies or benign tumors (e.g., papilloma, hemangioma)；
* Any intranasal and/or sinus surgery (including polypectomy) within 6 months prior to screening.
* Uncontrolled epistaxis within 2 months prior to screening.
* Regular use of decongestants (topical or systemic) prior to screening, except for short-term use during endoscopic examinations.
* Patients who have received any of the following treatments prior to randomization:

  * Treatment with immunosuppressants (including but not limited to: cyclophosphamide, cyclosporine, interferon gamma, azathioprine, methotrexate, mycophenolate, tacrolimus, Secukinumab) within 8 weeks or 5 half-lives prior to screening (whichever is longer)；
  * Treatment with any monoclonal antibodies (including but not limited to: benralizumab, mepolizumab, omalizumab, dupilumab, or other similar drugs [e.g., TSLP blockers]) within 8 weeks or 5 half-lives prior to screening (whichever is longer).
  * Patients who used medium- or short-acting systemic corticosteroids (SCS, including oral, intravenous, or intramuscular administration), systemic traditional Chinese medicine preparations for treating CRS within 4 weeks prior to screening, or received long-acting SCS (e.g., triamcinolone acetonide injection) within 6 weeks prior to screening, or who plan to receive the aforementioned medications during the study period.
  * Use of corticosteroid-eluting nasal stents within 6 months prior to screening;
  * Treatment with immunoglobulins or blood products within 28 days prior to screening;
  * Administration of live attenuated vaccines within 28 days prior to screening or planned during the study period;
  * Allergen-specific immunotherapy within 6 months prior to screening (allowed only if: initiated >3 months before screening, maintained at a stable dose for ≥1 month before Visit 1, and no planned dose changes during the study)；
  * Participation in other drug/medical device clinical trials within 3 months prior to screening (based on last administration/use).
  * Use nasal antihistamines (such as olopatadine nasal spray, azelastine nasal spray, levocabastine nasal spray, etc.) for the first 3 days.
* Screening for a history of active pulmonary tuberculosis within the past 12 months；
* Exclusion of infections within the last 14 days requiring systemic antibiotic, antiviral, antifungal, antiparasitic, or antiprotozoal therapy;
* Exclusion of subjects diagnosed with helminthic parasitic infection in the past 6 months who either did not receive standard treatment or had treatment failure；
* Known or suspected history of immunosuppression, immune dysfunction, or immune dysregulation, including but not limited to invasive opportunistic infections (histoplasmosis, listeriosis, coccidioidomycosis, pneumocystosis, aspergillosis), even if the infection has resolved; Or there is an unusual frequency, recurrence, or prolonged infection (as judged by the investigator).
* The forced expiratory volume in the first second (FEV1) of the subjects during the screening/introduction period was ≤ 50% of the normal predicted value.
* Patients with comorbid asthma who meet any of the following criteria:

Asthma exacerbation within 90 days before screening, or current use of inhaled corticosteroids (ICS) at a daily dose higher than 1000μg fluticasone (or equivalent).

Definition of Asthma Acute Exacerbation:

* Use of systemic corticosteroids (or a temporary increase in the stable dose of baseline OCS) for at least 3 consecutive days due to worsening asthma; a single injection of depot long-acting corticosteroids may be considered equivalent to a 3-day course of systemic corticosteroids.
* An emergency department or urgent care center visit due to asthma requiring systemic corticosteroids (as described above) (defined as evaluation and treatment in the emergency department or urgent care center lasting <24 hours).
* Hospitalization due to asthma (defined as admission to a medical facility and/or evaluation and treatment in a healthcare setting lasting ≥24 hours).

  * Use of leukotriene antagonists/modulators prior to randomization (subjects who have been on a stable dose of leukotriene modulators for ≥30 days continuously prior to randomization may be enrolled);
  * Presence of other concurrent active or clinically significant respiratory diseases that, in the investigator's judgment, may significantly impact the study, such as active tuberculosis, lung cancer, bronchiectasis, pulmonary sarcoidosis, pulmonary fibrosis, pulmonary hypertension, interstitial lung disease, or other active pulmonary conditions
  * Subjects who have undergone lobectomy or lung volume reduction surgery within 12 months prior to the start of the study;
  * Exclusion of subjects with cardiovascular conditions (including but not limited to unstable ischemic heart disease, heart failure, uncontrolled hypertension, myocardial infarction, significant arrhythmias, long QT syndrome, or Fridericia-corrected QT interval (QTcF) prolongation [≥450 ms in men, ≥470 ms in women]) if the investigator deems participation could compromise safety or study outcome interpretation;
  * Exclude individuals with difficult venous access or a history of vasovagal syncope (needle/blood-related);
  * Exclusion of any current active malignancy or history of malignancy (Patients with basal cell carcinoma, localized squamous cell carcinoma of the skin, or carcinoma in situ of the cervix are eligible if curative treatment was completed >12 months before V1. Patients with other malignancies are eligible if curative treatment was completed at least 5 years before V1).
  * Presence of active autoimmune diseases (including but not limited to Hashimoto's thyroiditis with hyperthyroidism, Graves' disease, inflammatory bowel disease, primary biliary cholangitis, systemic lupus erythematosus, multiple sclerosis and other neuroinflammatory disorders, psoriasis vulgaris, and rheumatoid arthritis);
  * Exclusion if any infectious disease screening indicator meets the following criteria during screening;
* Exclusion of subjects who are positive for hepatitis B virus surface antigen (HBsAg).
* Hepatitis B virus core antibody (HBcAb) with detectable Hepatitis B Virus (HBV)-DNA.
* Exclude if Hepatitis C Virus (HCV) antibody-positive and HCV-RNA positive, or if previously treated for HCV (regardless of current HCV-RNA status).
* Anti-Treponema pallidum antibody (Anti-TP) positive (if syphilis serology is positive, a non-treponemal test must be performed; subjects with a negative non-treponemal test and deemed by the investigator as previously cured are eligible).
* Anti-HIV positive

  * Abnormal laboratory test results:
* White blood cell count <3.5 × 10⁹/L;
* Aspartate aminotransferase (AST) >2.5 × upper limit of normal (ULN);
* Alanine aminotransferase (ALT) >2.5 × ULN;
* Total bilirubin >2 × ULN;
* Creatinine >1.5 × ULN

  * Any clinically significant abnormal findings during the import period, including physical examination, vital signs, 12-lead ECG, blood biochemistry, hematology, or urinalysis, which in the investigator's judgment may place the patient at risk, affect study results, or impair the patient's ability to complete the entire study
  * Women who are pregnant or lactating.
  * Those who were still smokers or had quit smoking for less than six months at the time of screening.
  * Exclude those with regular excessive alcohol consumption (>14 units/week for females or >21 units/week for males) in the past 6 months, inability to abstain during the trial, or a positive breath alcohol test.
  * History of drug abuse within the past 2 years, or a positive drug abuse screening result.
  * Subjects with a known history of hypersensitivity or allergic reaction to any ingredient of mometasone furoate nasal spray (Nasonex®) or TQC2731 injection.
  * Exclusion for any history of systemic allergic reaction to biologic agents (local injection site reactions excluded).
  * The participant demonstrated poor adherence and was deemed unable to complete the study.
  * Any medical or psychiatric condition that, in the judgment of the investigator or the sponsor's medical reviewer, may affect the subject's safety throughout the study or impede the subject's ability to complete the entire study process or interfere with the interpretation of study results, including but not limited to cardiovascular, gastrointestinal, hepatic, renal, neurological, musculoskeletal, infectious, endocrine, metabolic, hematologic disorders, psychiatric illnesses, or major physical disabilities.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Nasal Polyp Score (NPS) | From baseline to Week 24
  Change in Nasal Polyp Score (NPS) from baseline to Week 24 in CRSwNP subjects.
Nasal Congestion Score (NCS) | From baseline to Week 24
  Change in Nasal Congestion Score (NCS) from baseline to Week 24 in CRSwNP subjects
Change in nasal polyp score (NPS) from baseline | From baseline to Week 24
  Change in nasal polyp score (NPS) from baseline at week 24 in ECRSwNP subjects.
Change from baseline in Nasal Congestion Score (NCS) | From baseline to Week 24
  Change from baseline in Nasal Congestion Score (NCS) at Week 24 in ECRSwNP subjects

SECONDARY OUTCOMES:
Lund-Mackay score | From baseline to Week 24
  The change in Lund-Mackay score from baseline for the subject's CT scan at week 24. The higher the score, the more severe the CRS condition.
Olfactory loss score | From baseline to Week 60
  The change in anosmia score assessed in the electronic logs of subjects at each visit point relative to baseline. A reduction in the olfactory loss score implies therapeutic efficacy or ongoing recovery.
22-item Sino-Nasal Outcome Test (SNOT-22) score | From baseline to Week 60
  The change from baseline in the 22-item Sino-Nasal Outcome Test (SNOT-22) score at each visit.
Total Symptom Score (TSS) | From baseline to Week 60
  The change in Total Symptom Score (TSS) from baseline at each visit point for the subjects.
  A reduction in the Total Nasal Symptom Score (TSS) post-treatment suggests effective therapeutic response.
Visual Analog Scale (VAS) | From baseline to Week 60
  Visual Analog Scale (VAS) overall score changes for sinusitis relative to baseline at each visit point for subjects.
  A higher VAS score indicates a greater impact of sinusitis on the subject's quality of life.
The proportion of subjects receiving systemic corticosteroid (SCS) rescue or nasal polyp (NP) surgery | From baseline to Week 24
  The proportion of subjects receiving systemic corticosteroid (SCS) rescue or nasal polyp (NP) surgery during the 24-week double-blind treatment period
Time to systemic corticosteroid (SCS) rescue therapy or nasal polyp (NP) surgery | From baseline to Week 24
  Time to systemic corticosteroid (SCS) rescue therapy or nasal polyp (NP) surgery during the 24-week double-blind treatment period.
Numbers of participants with adverse events (AEs) and abnormal laboratory test results | From baseline until 30 days after the last dose
  Evaluate the safety of TQC2731 in subjects with CRSwNP, including abnormalities such as adverse events (AEs), laboratory tests, physical examinations, vital signs, and 12-lead electrocardiogram (ECG).
Incidence of anti-drug antibodies (ADA) | 2 hours pre-dose in Day 1, Day 57, Day 169, Day 253, Day 365, Day 421 and at the time of withdrawal
  Incidence of anti-drug antibodies (ADA)
Incidence of neutralizing antibodies (Nab) | 2 hours pre-dose in Day 1, Day 57, Day 169, Day 253, Day 365, Day 421 and at the time of withdrawal
  Incidence of neutralizing antibodies (Nab)
Blood eosinophil count | 2 hours pre-dose in Day 1, Day 169, Day 365, Day 421 and at the time of withdrawal
  Evaluate the changes from baseline in blood eosinophil count at each visit point.
Total Immunoglobulin E (IgE) concentration | 2 hours pre-dose in Day 1, Day 169, Day 365, Day 421 and at the time of withdrawal
  Evaluate the changes from baseline in peripheral blood total IgE at each visit point.
Nasal biopsy tissue eosinophil levels | 2 hours pre-dose in Day 1, Day 169, Day 365, Day 421 and at the time of withdrawal
  Evaluate the changes from baseline in nasal biopsy tissue eosinophil levels at each visit point.
Change in nonECRSwNP nasal polyp score (NPS) from baseline | From baseline to Week 24
  Change in nonECRSwNP nasal polyp score (NPS) from baseline at Week 24
The change from baseline in nonECRSwNP nasal congestion score (NCS) | Week 24
  The change from baseline in nonECRSwNP nasal congestion score (NCS) at week 24
The percentage of subjects with an NPS score improvement of ≥1 point from baseline | Baseline through week 60
  The percentage of subjects with an NPS score improvement of ≥1 point from baseline at each evaluation visit point.
The percentage of subjects with an NPS score improvement of ≥2 points from baseline | Baseline through week 60
  The percentage of subjects with an NPS score improvement of ≥2 points from baseline at each evaluation visit point.
The percentage of subjects with an improvement of ≥1 point in NCS score compared to baseline | Baseline through week 60
  The percentage of subjects with an improvement of ≥1 point in NCS score compared to baseline at each evaluation visit point.
The percentage of subjects with an improvement of ≥2 points in NCS score | Baseline through week 60
  The percentage of subjects with an improvement of ≥2 points in NCS score at each evaluation visit compared to baseline.

CONTACTS AND LOCATIONS:
Locations (60):
- China (60):
  - Zhongda Hosiptal Southeast University, Fuyang, Anhui
  - The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Peking University People'S Hospital, Beijing, Beijing Municipality
  - Beijing youan hospital，capital medical university, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The 940th Hospital of Joint Logistics Support force of Chinese People 's Liberation Army, Lanzhou, Gansu
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Second People'S Hospital, Shenzhen, Guangdong
  - Liuzhou People's Hospital, Liuchow, Guangxi
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Hebei Petro China Central Hospital, Langfang, Hebei
  - Hebei Medical University Third Hospital, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Hebei North University, Zhangjiakou, Hebei
  - Daqing People's Hospital, Daqing, Heilongjiang
  - Henan Provincial People'S Hospital, Zhengzhou, Henan
  - Jingzhou Central Hospital, Jingzhou, Hubei
  - Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - The First People's Hospital of Changde City, Changde, Hunan
  - People's Hospital of Hunan Province, Changsha, Hunan
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - Chifeng Municipal Hospital, Chifeng, Inner Mongolia
  - Affiliated Hospital of Inner Mongolia Medical University, Hohhot, Inner Mongolia
  - The First People'S Hospital of Lianyungang, Lianyungang, Jiangsu
  - Zhongda Hospital affiliated to Southeast University, Nanjing, Jiangsu
  - Jiangnan University Medical Center, Wuxi, Jiangsu
  - Xuzhou Medical University Affiliated Hospital, Xuzhou, Jiangsu
  - Affiliated Hospital of Yangzhou Univrtsity, Yangzhou, Jiangsu
  - Fengcheng People's Hospital, Fengcheng, Jiangxi
  - Ganzhou People's Hospital, Ganzhou, Jiangxi
  - The First Affiliated Hospital of NanChang University, Nanchang, Jiangxi
  - ShangRao People's Hospital, Shangrao, Jiangxi
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - The first hospital of Jilin University, Changchun, Jilin
  - Affiliated Zhongshan Hospital Of Dalian University, Dalian, Jilin
  - China Medical University Affiliated Shengjing Hospital, Shenyang, Liaoning
  - The Second Affiliated Hospital Of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The First Affiliated Hospital of Xi'an Jiao Tong University, Xi'an, Shaanxi
  - Yan'an University Xianyang Hospital, Xianyang, Shaanxi
  - Shandong Second Province General Hospital, Jinan, Shandong
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Zibo Central Hospital, Zibo, Shandong
  - Eye&ENT Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Zhongshan Hospital, Fudan University, Shanghai, Shanghai Municipality
  - Renji Hospital,Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai Sixth People's Hospital, Shanghai, Shanghai Municipality
  - Linfen Central Hospital, Lifen, Shanxi
  - First Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Yuncheng Central Hospital，Shanxi Province, Yuncheng, Shanxi
  - West China Hospital of Si chuan University, Chengdu, Sichuan
  - Chengdu Second People's Hospital, Chengdu, Sichuan
  - Tianjin First Central Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - Affilited hangzhou first people's hospital, school of medicine, westlakeuniversity, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Ningbo University, Ningbo, Zhejiang
  - Ningbo No.2 Hospital, Ningbo, Zhejiang
  - Taizhou First People's Hospital, Taizhou, Zhejiang